CLINICAL TRIAL: NCT01234558
Title: Randomized, Double Blind, Placebo Controlled, Single IV Dose Parallel Efficacy and Safety Study of GLYX-13 in Subjects With Inadequate/Partial Response to Antidepressants During the Current Episode of Major Depressive Disorder
Brief Title: Single IV Dose of GLYX-13 in Patients With Treatment-Resistant Depression
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Naurex, Inc, an affiliate of Allergan plc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GLYX13-C201
Record Dates: First submitted 2010-11-03; First posted 2010-11-04 (Estimated); Last update posted 2012-09-12 (Estimated); Status verified 2012-09

CONDITIONS: Major Depressive Disorder
Keywords: depression; NMDA antagonist; treatment resistant
MeSH Terms: conditions — Depressive Disorder, Major; Depression | interventions — GLYX-13 peptide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Normal Saline (Placebo Comparator): IV placebo
  Interventions: Drug: GLYX-13
- GLYX-13, 1 mg/kg (Experimental)
  Interventions: Drug: GLYX-13
- GLYX-13, 5 mg/kg (Experimental)
  Interventions: Drug: GLYX-13
- GLYX-13, 10 mg/kg (Experimental)
  Interventions: Drug: GLYX-13

INTERVENTIONS:
Drug: GLYX-13 — single IV dose
  Other Names: ThrProProThr

SUMMARY:
The purpose of this study is to determine whether GLYX-13 reduces depression score in patients with treatment-resistant depression.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of major depressive disorder consistent with DSM-IV-TR
* current episode greater than 8 weeks in duration
* Hamilton Depression score >/- 21
* less than 25% reduction in depression during current episode assessed by ATRQ

Exclusion Criteria:

* Axis diagnosis of other psychiatric disorders
* Experiencing hallucinations, delusions, other psychotic symptomatology
* ECT during current episode

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 115 (Actual)
Dates: Start 2011-05; Primary Completion 2012-06 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
Change in depression score | 14 days

SECONDARY OUTCOMES:
Change in BPRS+ | 14 days

CONTACTS AND LOCATIONS:
Overall Officials: Ronald M Burch, MD, PhD, Study Director — Naurex, Inc, an affiliate of Allergan plc; Vishaal Mehra, MD, Principal Investigator — Artemis Clinical Research, San Diego CA; Raymond Manning, MD, Principal Investigator — CNRI-LA, Pico Rivera CA; Paul Gross, MD, Principal Investigator — Lehigh Center for Clinical Research, Allentown PA; Surinder Randhawa, MD, Principal Investigator — Lynn Health Sciences Institute, Oklahoma City OK; David Greuner, MD, Principal Investigator — CRI-WW, Philadelphia PA; David Krefetz, DO, Principal Investigator — CRI-WW Lordes Hospital, Willingboro NJ; Benji Kurian, MD, Principal Investigator — U Texas SW Medical Center, Dallas TX; Michael Lesem, MD, Principal Investigator — Claghorn-Lesem Research Clinic, Houston TX; Matthew Macaluso, MD, Principal Investigator — Clinical Research Center, Univ Kansas, Wichita KS; Stephen Murray, MD PhD, Principal Investigator — Clinilabs, New York, NY
Locations (1):
- Mulitple, Evanston, Illinois, United States

REFERENCES:
- [Derived] Preskorn S, Macaluso M, Mehra DO, Zammit G, Moskal JR, Burch RM; GLYX-13 Clinical Study Group. Randomized proof of concept trial of GLYX-13, an N-methyl-D-aspartate receptor glycine site partial agonist, in major depressive disorder nonresponsive to a previous antidepressant agent. J Psychiatr Pract. 2015 Mar;21(2):140-9. doi: 10.1097/01.pra.0000462606.17725.93. PMID 25782764